CLINICAL TRIAL: NCT01758913
Title: Pharmacological Closure of Patent Ductus Arteriosus in Extreme Low Birth Weight Infants. A Comparison of Efficacy, Side Effects and Outcomes Between Indomethacin and Ibuprofen
Brief Title: Closure of Patent Ductus Arteriosus With Indomethacin or Ibuprofen in Extreme Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: Cook County Health (Other Government); China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDA Ind Ibu ELBW
Record Dates: First submitted 2012-12-16; First posted 2013-01-01 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Patent Ductus Arteriosus
Keywords: Bronchopulmonary dysplasia; patent ductus arteriosus; prostaglandin; Respiratory distress syndrome
MeSH Terms: conditions — Ductus Arteriosus, Patent; Bronchopulmonary Dysplasia; Respiratory Distress Syndrome | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibuprofen (Experimental): Infant who was assigned to ibuprofen, an initial dose of 10 mg/kg, followed by 5 mg/kg at 24 and 48 hours respectively as a course was given.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — To compare the efficacy, the side effects and the renal prostaglandin (PG) excretion between indomethacin and ibuprofen in extremely low birth weight (ELBW) infants.
  Other Names: 2-[4-(2-methylpropyl)phenyl]propanoic acid

SUMMARY:
Pharmacological closure of ductus arteriosus with prostaglandin (PG) inhibitors has been used for years. Previous studies indicated that ibuprofen has similar effect on ductal closure as indomethacin but has less adverse effects on renal function, cerebral blood flow and mesenteric blood flow.1-7 There are, however, very few studies being done specifically on extremely low birth weight (ELBW) infant < 1000 g. This group of infants has immature kidney and often has poor response to PG inhibitors and has high mortality and morbidity. We hypothesized that, in ELBW infants, the ductal and renal response to PG inhibitors may be different between indomethacin and ibuprofen.

DETAILED DESCRIPTION:
The aims of this study are to compare the efficacy, the side effects and the renal prostaglandin (PG) excretion between indomethacin and ibuprofen in extremely low birth weight (ELBW) infants. We enrolled one hundred and ten ELBW infants who had clinically significant and echo-evidence patent ductus arteriosus were assigned into 2 groups, 56 received indomethacin (0.2 mg/kg, 0.1 mg/kg and 0.1 mg/kg in 24 hours interval) and 54 received ibuprofen (10 mg/kg, 5mg/kg and 5 mg/kg in 24 hours interval). Serum electrolytes, creatinine, renal function (urine output, glomerular filtration rate (GFR), fractional excretion of sodium and potassium, osmolar clearance and free water clearance), urinary PG excretion, pulmonary outcome and mortality were all evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The selection criteria were: (1) preterm infants with birth weight <1000 g; 2) radiographic diagnosis of respiratory distress syndrome (RDS); (3) requirement of mechanical ventilation and (4) echocardiographic and clinical evidence of significant patent ductus arteriosus (PDA).

Exclusion Criteria:

* Exclusion criteria included: (1) evidence of infection or sepsis; 2) lethal congenital anomalies; (3) oliguria (< 1 ml/kg/h) and/or serum creatinine > 2.0 mg/dl and (4) low platelet count (< 50,000/mm3) or bleeding tendency.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2007-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of infants with ductus closure | 6 months
  To compare the number of infants with ductus closure treated with indomethacin and ibuprofen in extremely low birth weight infants.

SECONDARY OUTCOMES:
Urine output | 1 month
  To compare the urine output between indomethacin and ibuprofen treatment in extremely low birth weight infants.

OTHER OUTCOMES:
Serum creatinine | 1 month
  To compare serum creatinine between indomethacin and ibuprofen treatment in extremely low birth weight infants.

CONTACTS AND LOCATIONS:
Overall Officials: Tsu-Fu Yeh, MD, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois, United States

REFERENCES:
- [Background] Yeh TF, Achanti B, Patel H, Pildes RS. Indomethacin therapy in premature infants with patent ductus arteriosus--determination of therapeutic plasma levels. Dev Pharmacol Ther. 1989;12(4):169-78. PMID 2766920
- [Background] Yeh TF, Raval D, Luken J, Thalji A, Lilien L, Pildes RS. Clinical evaluation of premature infants with patent ductus arteriosus: a scoring system with echocardiogram, acid-base, and blood gas correlations. Crit Care Med. 1981 Sep;9(9):655-7. doi: 10.1097/00003246-198109000-00009. PMID 7273813
- [Background] Yeh TF, Luken J, Raval D, Thalji A, Carr I, Pildes RS. Indomethacin treatment in small versus large premature infants with ductus arteriosus. Comparison of plasma indomethacin concentration and clinical response. Br Heart J. 1983 Jul;50(1):27-30. doi: 10.1136/hrt.50.1.27. PMID 6860508